CLINICAL TRIAL: NCT02878213
Title: DURABLE-I Study: Dielectric Unravelling of Radiofrequency ABLation Effectiveness
Acronym: DURABLE-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-D700-004
Record Dates: First submitted 2016-07-28; First posted 2016-08-25 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D700 System (Experimental): Patients referred to catheter-based Atrial-Fibrillation (AF) ablation procedure therapy comprising of Pulmonary Veins Isolation (PVI).
  Interventions: Device: D700 System

INTERVENTIONS:
Device: D700 System — Atrial Fibrillation Ablation Procedure

SUMMARY:
The purpose of this study is to evaluate real-time gap detection using EPD D700 dielectric sensing compared with customary electrical isolation tests and Adenosine infusion at the end of the procedure. Furthermore, safety, usability and clinical applicability of the system for guided AF ablation will be confirmed.

DETAILED DESCRIPTION:
Prospective, single-center, non-randomized, non-blinded, open label, and single arm study.

All procedures will be performed under CARTO-3 guidance for the treatment of atrial fibrillation (AF). The EPD D700 system will be used in-tandem, to record pre-, during and immediate post-ablation tissue characteristics and compute likelihood of lesion transmurality and permanency. Additionally, D700 system safety, feasibility, usability and clinical applicability will be documented.

The entire procedure will be conducted as customary, using standard and approved off-the-shelf equipment (body surface electrodes, diagnostic and irrigated ablation catheters, RF generator and recording system), in a completely clinically independent manner from the EPD D700 system. The physician will neither use nor rely on any of the D700 system output for clinical decision making and will be blinded to the D700 lesion assessment forecasts. After 30 days following the initial procedure, a repeated procedure will be performed for gap detection and its results will be correlated with the D700 predictions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age ≥ 18 and ≤ 80 years.
2. Paroxysmal atrial fibrillation (PAF)
3. Able to provide written informed consent form to participate in the study, prior to any study related procedures.
4. Able and willing to comply with the study protocol requirements.
5. A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days.

Exclusion Criteria:

1. Any planned surgical or endovascular intervention within 30 days before or after the index procedures.
2. Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint.
3. Previous AF ablation therapy.
4. Clinical evidence of active coronary ischemia, significant Valvular heart disease, or hemodynamically significant congenital cardiac abnormality.
5. Patient had experienced myocardial infarction (MI), stroke (CVA) or transient ischemic attack (TIA) or other neurological disturbances.
6. Patient has a pacemaker.
7. Thrombi detected in the heart.
8. Life expectancy less than 12 months.
9. Known severe renal insufficiency.
10. Known allergy to Iodine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- Arrhythmia Department and Electrophysiology Laboratory, State Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For DURABLE-1 22 consecutive paroxysmal atrial fibrillation patients were recruited.
  The trial was extended (DURABLE-1.1) and altogether 39 paroxysmal atrial fibrillation patients were recruited.
Groups:
- D700 (KODEX-EPD) System: Paroxysmal Atrial Fibrillation (PAF) patients referred to catheter-based Atrial-Fibrillation (AF) ablation procedure therapy comprising of Pulmonary Veins Isolation (PVI).
  D700 (KODEX-EPD) System: Atrial Fibrillation Ablation Procedure
Period: Overall Study
Arm/Group | D700 (KODEX-EPD) System
Started | 39
Completed | 36
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | D700 System
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 36
Arterial Hypertension [Number; unit: participants] | 25
Diabetes Mellitus [Count of Participants; unit: Participants] | 5
Valvular Heart Disease [Count of Participants; unit: Participants] — Moderate Mitral Regurgitation
  Participants | 5
Moderate Alcohol Consumption [Count of Participants; unit: Participants] | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.15 (5.4)
NSR during procedure [Count of Participants; unit: Participants] | 31
NYHA functional class [Mean (Standard Deviation); unit: class] — NYHA Functional Classification
  1-Mild-Patients with cardiac disease but without resulting in limitation of physical activity. 2-Mild-Patients with cardiac disease resulting in slight limitation of physical activity.
  3-Moderate-Patients with cardiac disease resulting in marked limitation of physical activity.
  4-Severe-Patients with cardiac disease resulting in the inability to carry on any physical activity without discomfort.
  class | 1.7 (1.1)
CHAD2 [Mean (Full Range); unit: units on a scale] — The CHA₂DS₂-VASc value is clinical prediction rules for estimating the risk of stroke in patients with non-rheumatic atrial fibrillation.
  Risk Factor (Letter) and Score (Number):
  C - Congestive heart failure (1) H - Hypertension (1) A - Age ≥75 years (2) D - Diabetes Mellitus (1) S - Prior Stroke or TIA (2) V - Vascular disease (1) A - Age 65-74 years (1) Sc - Sex category (female) (1)
  Maximum value is the total sum of the risks numbers, which is 10. Minimum value will be only one risk which is 1.
  units on a scale | 1.8 [1 to 10]
Diagnosis to ablation time [Mean (Standard Deviation); unit: months] | 46 (33)
LA diameter [Mean (Standard Deviation); unit: cm] | 5.2 (0.7)
LAA morphology [Count of Participants; unit: Participants]
  Cauliflower | 16
  Chicken wing | 12
  Windsock | 5
  Cactus | 3

OUTCOME MEASURES:

1. Primary Outcome: ETA Reading at Index Procedure vs. Actual Gaps at 1-month Restudy
Description: ETA Reading at Index Procedure vs. Actual Gaps at 1-month Restudy. All patients underwent PVI at index procedure. The physicians were blinded to the D700 (KODEX-EPD) ETA function pairwise real-time lesion assessment readings.
  All patients were restudied at 1-mont, and ETA reading, which is the number of gaps as predicted by the system, were compared to the actual gaps as validated in the second procedure after one month.
Time Frame: 30 days
Population: Analyzed ablation pairs in all participants
Measure: Number; unit: participants
Groups:
- D700 (KODEX-EPD): ETA Reading at Index Procedure vs. Actual Gaps at 1-month Restudy in all patients
Arm/Group | D700 (KODEX-EPD)
Number analyzed (Participants) | 36
participants
  No 1-month gaps: Positive ETA reading at index | 231
  No 1-month gaps: Negative ETA reading at index | 1549
  Actual 1-month gaps: Positive ETA reading at index | 48
  Actual 1-month gaps: Negative ETA reading at index | 13

2. Primary Outcome: 1-month Patient Analysis
Description: ETA Reading at Index Procedure vs. Actual Gaps at 1-month Restudy
Time Frame: 30 days
Population: All patients were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- D700 (KODEX-EPD): All patients in which the KODEX-EPD system was used.
Arm/Group | D700 (KODEX-EPD)
Number analyzed (Participants) | 36
Participants
  1-month gaps: number analyzed (Participants) | 27
  1-month gaps: Positive ETA reading at index procedure | 18
  1-month gaps: Negative ETA reading at index procedure | 9
  No 1-month gaps: number analyzed (Participants) | 9
  No 1-month gaps: Positive ETA reading at index procedure | 9
  No 1-month gaps: Negative ETA reading at index procedure | 0

ADVERSE EVENTS:
Time Frame: 1 month; Hospitalization periods - index procedure and restudy (after 1 month from the first procedure), until discharge;
Groups:
- D700 (KODEX-EPD): All patients in which the KODEX-EPD system was used included in the group.
Arm/Group | D700 (KODEX-EPD)
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D700 (KODEX-EPD) (N=39)
TIA (Nervous system disorders) | 1 (1) — The patient has developed signs of stroke following transseptal before cardiac mapping of the left atrium was initiated. The procedure was immediately aborted. All neurological deficits have resolved within a few days while in hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT02878213/Prot_SAP_000.pdf